CLINICAL TRIAL: NCT04258423
Title: Preservation of Renal Function After Liver Transplant for Patients With Pre-existing Chronic Kidney Disease or Peri-operative Acute Kidney Injury Using Everolimus Plus Mycophenolate Mofetil Immunosuppression Regimen
Brief Title: Everolimus Plus Mycophenolic Acid for Kidney Preservation in Liver Transplant Recipients With Impaired Kidney Function
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was larger than expected and became a burden to faculty and staff resources.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chandrashekhar Kubal, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1807596072
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Intervention Model Description: Tacrolimus as maintenance immunosuppression, then randomized to Everolimus plus Mycophenolate Mofetil, discontinuing Tacrolimus once Everolimus level within goal range OR randomized to continued maintenance with Tacrolimus plus Mycophenolate Mofetil.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Tacrolimus as maintenance immunosuppression
  Interventions: Drug: Tacrolimus
- Study Arm (Experimental): Everolimus as maintenance immunosuppression
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Tacrolimus — Low dose Tacrolimus
  Other Names: Prograf
  Arms: Control Arm
Drug: Everolimus — Everolimus
  Other Names: Zortress
  Arms: Study Arm

SUMMARY:
Tacrolimus is the standard immunosuppressive drug used to prevent organ rejection post liver transplant. One side effect of Tacrolimus is nephrotoxicity. Everolimus does not have the nephrotoxicity side effects of Tacrolimus. Replacement of Tacrolimus by Everolimus may have a reduced incidence of renal dysfunction in liver transplant patients who already have chronic kidney disease or peri-operative acute kidney injury. Liver transplant patients receive potent induction immunosuppression in the form of rabbit anti thymocyte globulin. Investigators believe that in conjunction with this induction regimen, patients can be maintained on Everolimus monotherapy without the risk of rejection. Additionally, Everolimus is known to induce tolerance in transplant recipients. Tolerant patients do not require immunosuppression to accept transplant organs. Tacrolimus is a widely used in liver transplant recipients for immunosuppression, however it is associated with nephrotoxicity. Everolimus, on the other hand lacks nephrotoxicity. Whether replacement of tacrolimus by Everolimus preserves kidney function in patients with pre-existing chronic kidney disease or acute kidney injury is not well established. Also, the efficacy and safety of reduced-dose Everolimus with or without Mycophenolate Mofetil in prevention of rejection is unknown.

Primary Aim Assess the effect of Everolimus with or without Mycophenolate Mofetil versus Tacrolimus plus Mycophenolate Mofetil therapy on renal function measured by Glomerular Filtration Rate (GFR). Secondary Aims

Compare the efficacy of Everolimus plus Mycophenolate Mofetil versus Tacrolimus plus Mycophenolate Mofetil therapy as measured by the following:

* Biopsy-confirmed acute rejection
* Hyperlipidemia
* Proteinuria
* % regulatory T-cells in circulation
* NODAT [New Onset Diabetes mellitus After Transplant], hypertension and malignancy
* Tolerance measured by gene profiling at year 1, 2 and 3

DETAILED DESCRIPTION:
Following transplant, prior to the one month post transplant visit, subjects will be approached either in the transplant unit in the hospital or at the transplant clinic in the hospital for study participation. Following enrollment, subjects will be randomized at one month post transplant to reduced dose Tacrolimus plus Mycophenolate Mofetil immunosuppression (control group) or to Everolimus plus Mycophenolate Mofetil (study group) maintenance immunosuppression.

After liver transplant, all patients will receive the standard induction regimen and Tacrolimus monotherapy.

INDUCTION:

Rabbit anti-thymocyte globulin (rATG) 1.5 mg/kg of actual body weight rounded to nearest 25 mg and capped at 150 mg for up to three doses given IV on post-operative day (POD) 1, 3, and 5. Some patients may receive only one dose if considered too frail to need all three doses.

30 minutes prior to infusion, pre-medicate with the following: Daily steroid dose Acetaminophen (Tylenol®) 650 mg PO or per NG x 1 dose B - Lay Summary & Research Design Diphenhydramine (Benadryl®) 25 mg IV push x 1 dose

Steroids:

Methylprednisolone (Solu-Medrol®) 250 mg IV push x 1 dose on POD 1 (given 30 minutes prior to rATG) and 125 mg IV push x 1 dose on POD 3.

Maintenance:

Low dose Tacrolimus (FK / Prograf®) (titrated to a goal trough of 6 ± 1 ng/mL) plus Mycophenolate Mofetil 500 mg BID.

RANDOMIZATION:

On POD 30, patients meeting study criteria will be randomized to either the study arm or control arm. Patients randomized to the study arm will be converted to Everolimus (target trough levels 4-8 ng/mL) plus Mycophenolate Mofetil 500 mg BID therapy. The control arm will be maintained on the low dose Tacrolimus plus Mycophenolate Mofetil therapy.

At 3 months, patients with GFR <=60 will proceed to reduced dose Everolimus (target trough levels 3-6 ng/mL) plus Mycophenolate Mofetil 500 mg BID therapy. Patients with GFR >60 will proceed to Everolimus monotherapy (target trough levels 4-8 ng/mL).

Complete blood counts, liver function panels, and drug levels will be monitored per Standard of Care [SOC]: initially twice per week for first month, once per week for next two months, once every other week for next three weeks, and then once monthly. Ultrasound, ERCP, biopsy as needed by clinical situation as SOC.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipients ≥ 18 years old
* Baseline renal dysfunction (GFR ≤ 60 mL/min)
* Rabbit anti-thymocyte globulin (rATG) induction (cumulative dose 3 - 5 mg/kg)
* Indication for transplant: ethanol, hepatitis C, or nonalcoholic steatohepatitis

Exclusion Criteria:

* Increased risk of rejection: autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, positive crossmatch, retransplantation
* Incompletely healed incision or other wound healing issues at time of randomization
* Multiple or previous organ transplantation
* Severe, uncontrolled hypercholesterolemia (> 9mmol/L) or hypertriglyceridemia (>8.5 mmol/L) in the 6 mo prior to transplantation
* Insurance company unwilling to pay for the cost of the everolimus
* Pregnant women
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandrashekhar Kubal, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Tacrolimus as maintenance immunosuppression
  Tacrolimus:
  Low dose Tacrolimus (FK / Prograf®) (titrated to a goal trough of 5 ± 1 ng/mL)
- Study Arm: Everolimus as maintenance immunosuppression
  Everolimus: Everolimus (target trough levels 4-8 ng/mL) initiated at 1mg BID. Tacrolimus will be discontinued once Everolimus level is within goal or at the discretion of the provider
Period: Overall Study
Arm/Group | Control Arm | Study Arm
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study Closure | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Study Arm | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 60 [59 to 61] | 61 [58 to 64] | 60.5 [58 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate in Patients Treated With Tacrolimus
Description: Glomerular Filtration Rate
Time Frame: 36 months post-transplant
Population: Study was terminated prior to any subject reaching the 36 Month timepoint. No data were collected for this outcome measure.
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Glomerular Filtration Rate in Patients Treated With Everolimus
Description: Glomerular Filtration Rate
Time Frame: 36 months post-transplant
Population: as for outcome 1
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Patients Who Experience Transplant Rejection
Description: Biopsy
Time Frame: 36 months post-transplant
Population: as for outcome 1
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Control Arm | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=2) | Study Arm (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Pt has history of anemia prior to transplant. He has several infusions since transplant. Was admitted to ED for transfusion and observation following reading of 6.4 g/dL. He was discharged same day and has been trending around 8.8 d/dL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT04258423/Prot_SAP_000.pdf